CLINICAL TRIAL: NCT05144880
Title: Effects of Electroacupuncture With Different Frequencies for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Li, Attending Doctor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020YKJ08
Record Dates: First submitted 2021-11-14; First posted 2021-12-03 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture with 2Hz group (Experimental)
  Interventions: Other: electroacupuncture
- electroacupuncture with 100Hz group (Experimental)
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — A total of 12 treatment sessions will be administered to each participant. The acupoints of needles inserted for each participant in each session are DU20, EX-HN1, DU29, HT17, PC6, RN6, RN4, LR3 and SP6. The needles will be manually stimulated by rotating, thrusting, stirring, etc. to produce ''De Qi'' sensation. Then we will use electroacupuncture for acupoint stimulation lasting 30min. The frequency will be set as 2Hz for the electroacupuncture with 2Hz group and the frequency will be set as 100Hz for the electroacupuncture with 100Hz group.

SUMMARY:
Two groups of subjects will be included 55 subjects in electroacupuncture with 2Hz group, 55 subjects in the electroacupuncture with 100Hz group. The clinical efficacy of electroacupuncture with different frequencies (2 Hz, 100 Hz) in the treatment of MDD will be observed by evaluation indicators, such as Self-rating depression scale and Hamilton depression scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suﬀering from MDD in accordance with the diagnostic criteria;
2. Hamilton Depression Scale score is between 21 and 35 (mild to moderate MDD);
3. 18≤age≤60 years, both gender;
4. Patients who have not used antidepressants and other psychiatric drugs (including traditional Chinese medicine), or have used them but have stopped for at least 2 weeks;
5. Patients have clear consciousness and could communicate with others normally;
6. Patients could understand the full study protocol and written informed consent is provided by themselves. Note: Subjects who meet the above six items will be included.

Exclusion Criteria:

1. Patients with bipolar disorder;
2. Patients with schizophrenia or other mental disorders;
3. Patients with severe medical diseases, tumors or diseases of the central nervous system;
4. Patients suﬀering from severe depressive episode with psychotic symptoms;
5. Suicidal patients;
6. Patients with seasonal depression;
7. Patients with organic depression;
8. Patients with alcohol or drug addicts;
9. Patients using other therapies;
10. Patients in pregnancy or lactation;
11. Patients suffering from cognitive dysfunction, aphasia or other diseases that cannot cooperate with treatment;
12. Patients with pacemakers;
13. Patients who are not suitable for electroacupuncture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety and depression severity measure by Self-rating depression scale（SDS） | There will be evaluated before intervention, at 2, 4weeks after intervention and at the end of 4-weeks follow-up.
  This scale contains 20 items that reflect the subjective feelings of depression, 10 of which are positive scores and 10 are reverse scores. Each item is divided into four grades according to the frequency of symptoms, If it is a positive scoring question, it will be rated as 1, 2, 3, and 4 points; for a reverse scoring question, it will be rated as 4, 3, 2, and 1. After the evaluation, add up the scores in the 20 items to get the total rough score, and then multiply the rough score by 1.25 and take the integer part to get the standard score
Change in the severity of depression measure by Hamilton depression scale (HAMD) | There will be evaluated before intervention, at 2, 4weeks after intervention and at the end of 4-weeks follow-up.
  This scale is performed by two trained raters to perform a HAMD, usually in the form of conversation and observation. After the examination, the two raters will score independently

SECONDARY OUTCOMES:
Change in sleep quality measured by Insomnia severity index (ISI) | There will be evaluated before intervention, at 2, 4weeks after intervention and at the end of 4-weeks follow-up.
Change in Traditional Chinese medicine syndrome score | There will be evaluated before intervention, at 2, 4weeks after intervention and at the end of 4-weeks follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaoyu Li, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR